CLINICAL TRIAL: NCT02929979
Title: Cognitive Remediation for Alcohol Use Disorder and Posttraumatic Stress Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: D1492-W; 1IK2RX001492-01A1 (NIH)
Record Dates: First submitted 2016-09-28; First posted 2016-10-11 (Estimated); Results first posted 2021-02-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-01

CONDITIONS: Alcohol Use Disorder; PTSD; Cognitive Dysfunction
Keywords: PTSD; Alcohol Use Disorder; Cognitive Training; Veterans
MeSH Terms: conditions — Alcoholism; Stress Disorders, Post-Traumatic; Cognitive Dysfunction | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive Training (Experimental): Participants will complete 22.5 hours of cognitive training exercises over 6-weeks (training 5 times a week) using an app-based program, BrainHQ. BrainHQ is based on a previous neuroscience-based cognitive training program shown to improve cognition in several different randomized controlled studies with other clinical populations. The investigators will use a suite of BrainHQ exercises designed to target and ameliorate cognitive disruptions in 4 cognitive domains (see main outcome). The investigators will employ basic exercises that focus on increasing processing efficiency in the auditory and visual perceptual and working memory domains, as well as exercises that target impulsivity and cognitive biases. Exercises will be packaged into 4 modules (attention skills, memory skills, executive functioning skills, cognitive control skills) comprised of 4 exercises each. All participants will progress through the same fixed schedule of modules.
  Interventions: Behavioral: Cognitive Training
- Placebo control (Placebo Comparator): Participants will play a rotating set of commercial computer games at the same dose and frequency as the cognitive training. The investigators selected this control activity because it mirrors the game-like properties of the cognitive training and it will be used to control for contact with research personnel and for the non-specific effects of participant motivation and engagement with daily computerized activities. It also allows for a double blind study design. Games from the website Sporcle will be used and an online account can be created for each participant.
  Interventions: Behavioral: Cognitive training placebo control

INTERVENTIONS:
Behavioral: Cognitive Training — Participants will complete 22.5 hours of cognitive training exercises over 6-weeks (training 5 times a week) using an app-based program, BrainHQ (BPI/Posit Science, San Francisco). BrainHQ is based on a previous neuroscience-based cognitive training program shown to improve cognition in several different randomized controlled studies with other clinical populations. The investigators will use a suite of BrainHQ exercises designed to target and ameliorate cognitive disruptions in 4 cognitive domains (see main outcome). The investigators will employ basic exercises that focus on increasing processing efficiency in the auditory and visual perceptual and working memory domains, as well as exercises that target impulsivity and cognitive biases. Exercises will be packaged into 4 modules (attention skills, memory skills, executive functioning skills, cognitive control skills) comprised of 4 exercises each. All participants will progress through the same fixed schedule of modules.
  Arms: Cognitive Training
Behavioral: Cognitive training placebo control — Participants will play a rotating set of commercial computer games at the same dose and frequency as the cognitive training. The investigators selected this control activity because it mirrors the game-like properties of the cognitive training and it will be used to control for contact with research personnel and for the non-specific effects of participant motivation and engagement with daily computerized activities. It also allows for a double blind study design. Games from the website Sporcle will be used and an online account can be created for each participant.
  Arms: Placebo control

SUMMARY:
The project will examine whether a computerized neuroscience-based cognitive training program can improve cognitive functioning and recovery outcomes among Veterans with Alcohol Use Disorder and co-occurring PTSD. Information from this study will help determine the malleability of cognitive dysfunction, an established risk factor for poor recovery outcomes in this population. Improved functional outcomes can decrease risk of chronic impairment and ultimately help affected individuals live richer, more productive lives. Web-based treatment technologies may increase the reach and impact of treatment, and foster patient recovery in cases where staffing, space, acceptability of counseling, and transportation are barriers. Findings may also support expanding use of existing, highly-accessible cognitive remediation technologies to other vulnerable clinical populations.

DETAILED DESCRIPTION:
The prevalence of Alcohol Use Disorder (AUD), Posttraumatic Stress Disorder (PTSD) and co-occurring AUD and PTSD is elevated among Veterans compared to civilians (Carter et al., 2011). Despite available empirically supported treatments, relapse and non-response rates remain high and individuals with co-occurring AUD and PTSD evidence particularly poor clinical and functional outcomes (McCarthy & Petrakis, 2010). Given recent estimates that 63-76% of Operation Enduring Freedom/Operation Iraqi Freedom (OEF/OIF) Veterans with an AUD also have a diagnosis of PTSD (Seal et al., 2011), there is urgent need to reduce chronic impairment among this growing and highly vulnerable population.

AUD and PTSD are characterized by separate and overlapping deficits in attention, memory and higher-order skills known as executive functions (e.g., planning, inhibition, self-regulation), which are in turn, associated with poor clinical and functional outcomes (Bates et al., 2013; Polak et al., 2012, Aupperle, 2012). Indeed, cognitive dysfunction can interfere with many aspects of recovery (e.g. gaining control of maladaptive, over-trained behaviors) and its targeting as a trans-disease process for direct intervention represents a potentially high-yield and innovative approach for optimizing recovery outcomes. Neuroscience-based computerized cognitive training programs for psychiatric illness have achieved growing support in the literature and demonstrate strong potential to remediate disrupted cognitive processes observed in AUD and co-occurring PTSD (Bates et. 2013; Vinogradov et al., 2012). These programs offer a highly accessible, individualized, patient-driven, non-medication treatment approach for improving cognitive functioning. Such improvements may increase emotional and behavioral control and enhance patients' capacity to effectively employ more adaptive self-management strategies. To date however, no studies have capitalized on available evidence-based cognitive remediation technologies to comprehensively target patterns of neurocognitive dysfunction that underlie both AUD and PTSD.

The proposed Rehabilitation Research and Development (RR&D) Career Development Award-2 (CDA-2) seeks to fill this gap by conducting a randomized prospective study, designed to evaluate the feasibility and efficacy of an existing web-based cognitive training program (BrainHQ; Posit Science/Brain Plasticity Institute) versus a placebo, for improving cognitive functioning and recovery outcomes. The research will be conducted iteratively, in two stages, based on the Stage Model of Behavioral Therapy Development per the National Institute on Drug Abuse, and has two overarching aims: Aim 1: Examine the acceptability, usability and feasibility of an existing web-based cognitive training program tailored for AUD and co-occurring PTSD. Aim 2: Test the efficacy of the web-based cognitive training program to improve cognitive functioning as well as clinical and functional outcomes. To test these aims, 148 Veterans with AUD and PTSD will be recruited from an outpatient Substance Use Disorder (SUD) treatment program. Participants will be randomized into either cognitive training or a computer game control. Individuals will then complete a baseline assessment, followed by 30 hours of home-based cognitive training or computer games over 6 weeks. Assessments will be completed each week of the training, as well as post-training and at post-training follow-up. The primary outcome will be performance on an (untrained) neuropsychological assessment battery 6 months post-training. Secondary outcomes include alcohol use, PTSD symptoms and quality of life.

Findings from the proposed study will inform clinical practice and policy by investigating whether a cognitive training program (shown to improve cognitive functioning in other clinical populations) can improve cognitive functioning and promote gains in functional recovery from AUD and PTSD. This study will lay the groundwork to investigate the potential for cognitive training to remediate neurocognitive disruptions in other dually diagnosed SUD patient populations across different VA treatment programs. This translational program of research will help vulnerable Veteran populations achieve more optimal and enduring recovery outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Be a Veteran
* Meet DSM-5 diagnostic criteria for current AUD
* Meet DSM-5 criteria for current PTSD
* Be willing to perform daily home-based computer exercises for 6 weeks

Exclusion Criteria:

Individuals will be excluded based on evidence of the following:

* History of, or current, psychotic disorder or Schizophrenia
* Current scheduled (i.e., daily) prescribed use of cognitive enhancers (e.g., Memantine) or stimulants (e.g., Methylphenidate) that may enhance cognitive performance
* Current severe traumatic brain injury (DoD TBI Screen 2)
* Any type of dementia (Mini Mental Status Exam (MMSE) < 24), delirium or medical illnesses associated with potential cognitive issues (HIV, Hypothyroidism, B-12 deficiency)
* Any level of mental retardation (Wechsler Test of Adult Reading WTAR)
* Limited ability to speak/read/write/understand English (WTAR)
* Inadequate vision or hearing
* Active suicidal/homicidal intent
* Self-report and collateral history from medical record/primary care physician/outpatient addiction treatment team will be used as necessary to determine inclusion and exclusion.

  * Suicidal and homicidal intent will be assessed in the context of a structured clinical interview.
  * In the unlikely event that respondents endorse active intent they will be referred immediately for treatment and will be excluded from the current study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-07-21 (Actual); Study Completion 2019-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrienne Julie Heinz, PhD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sporcle Website — http://www.sporcle.com
- See also: The Iowa Gambling Task — https://idp.springer.com/authorize/casa?redirect_uri=https://link.springer.com/content/pdf/10.1007/s11065-009-9083-4.pdf&casa_token=leCw-mNAgLIAAAAA:8srfkEu1hKO2QF2wJPOvXb2bmZrTBh2VWQN_8AtdKA8z7v2LKW1TlNz_SZcUYySBCeZLSrkr2Tnw7Ti8Hg

RESULTS

PARTICIPANT FLOW:
Groups:
- Cognitive Training: Participants will complete 22.5 hours of cognitive training exercises over 6-weeks (training 5 times a week) using an app-based program, BrainHQ. BrainHQ is based on a previous neuroscience-based cognitive training program shown to improve cognition in several different randomized controlled studies with other clinical populations.
- Placebo Control: Participants will play a rotating set of commercial computer games at the same dose and frequency as the cognitive training. Games from the website Sporcle were used for each participant.
Period: Overall Study
Arm/Group | Cognitive Training | Placebo Control
Started | 52 | 38
Completed | 25 | 28
Not Completed | 27 | 10

BASELINE CHARACTERISTICS:
Population: full sample that entered intervention
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Training | Placebo Control | Total
Number analyzed (Participants) | 52 | 38 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.41 (11.43) | 40.41 (11.43) | 40.41 (11.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 48 | 35 | 83
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 6 | 15
  Not Hispanic or Latino | 43 | 32 | 75
  Unknown or Not Reported | 0 | 0 | 0
Posttraumatic Stress Disorder [Count of Participants; unit: Participants] | 52 | 38 | 90

OUTCOME MEASURES:

1. Primary Outcome: The Revised Hopkins Verbal Learning Test
Description: The Revised Hopkins Verbal Learning Test (HVLT-R; Brandt & Benedict, 2001) assesses learning and memory for a 12-word list (organized into three semantic categories) immediately after the list is read (trial 1), cumulatively across trials (sum trials 1-3) and after a delay (free recall after 25 minutes). Test scores were normalized to t-scores with a Test mean = 50; SD =10 and higher scores indicate better verbal learning and memory.
Time Frame: 6-weeks
Population: t-test; data were missing for some participants due to attrition
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo Control: Cognitive training placebo control: Participants will play a rotating set of commercial computer games at the same dose and frequency as the cognitive training. The investigators selected this control activity because it mirrors the game-like properties of the cognitive training and it will be used to control for contact with research personnel and for the non-specific effects of participant motivation and engagement wi
Arm/Group | Cognitive Training | Placebo Control
Number analyzed (Participants) | 21 | 22
units on a scale | 47.71 (10.34) | 44.14 (10.70)

2. Primary Outcome: The Wechsler Adult Intelligence Scale-IV Working Memory Index
Description: The Wechsler Adult Intelligence Scale-IV (WAIS-IV; Wechsler, 2008) Working Memory Index subtests will be employed: (1) Digit Span - participants are asked to repeat a number sequence, repeat in reverse order and then repeat in a sequential order; (2) Arithmetic - participants are asked to mentally solve arithmetic word problems within a time limit; (3) Letter-Number Sequencing - participants are asked to recall a combination of numbers and letters that they must first numerically and alphabetically sequence. Test scores are standardized on a normed scale with a Test mean = 100; SD =15 and higher scores indicate better working memory.
Time Frame: 6-weeks
Population: t-test; some data were missing due to attrition
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Training | Placebo Control
Number analyzed (Participants) | 21 | 22
units on a scale | 102 (14.34) | 103.27 (13.99)

3. Primary Outcome: The Conners' Continuous Performance Task II
Description: The Conners' Continuous Performance Task II (CPT-II; Conners & Staff, 2000) is a computerized task that assesses vigilance and sustained attention. The participant is presented with a stimulus at variable interstimulus event rates and is asked to respond to all stimuli except the "X." Thus they must maintain a continuous response set (sustained attention) and inhibit responding when a specific target is presented. Test scores are normed on a t-score with a Test mean = 50; SD =10; higher scores indicate better response inhibition.
Time Frame: 6-weeks
Population: t-test; missing data for some participants due to attrition or technical difficulties in test administration
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Training | Placebo Control
Number analyzed (Participants) | 26 | 28
units on a scale | 47.92 (10.59) | 50.11 (8.44)

4. Primary Outcome: The Color-Word Interference Test (DKEFS)
Description: The Color-Word Interference Test is included in the DKEFS tests (DKEFS; Delis, Kaplan, & Kramer, 2001) and is a variant of the Stroop procedure. Participants are asked to name the ink color (e.g., blue) in which different color words (e.g., red) are printed and thus the test captures ability to inhibit an overlearned response. Test scores are normed on a standardized scale with a Test mean = 10; SD = 3; higher scores indicate better response inhibition.
Time Frame: 6-weeks
Population: t-test; missing data for some participants due to attrition or technical difficulties in test administration
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Training | Placebo Control
Number analyzed (Participants) | 21 | 22
units on a scale | 10.86 (2.37) | 10.55 (2.20)

5. Primary Outcome: The Iowa Gambling Task
Description: The Iowa Gambling Task (IGT; Bechara et al., 1994) is computerized and participants select from among 4 decks of cards that vary in monetary reward and punishment (i.e., risky "bad" decks that result in infrequent but large losses and "good" decks that result in gradual monetary gain over repeated trials). The IGT will be used to assess decision-making. Money earned is the primary outcome with more money earned indicated better decision making. Go to the links in the Reference section to learn more about this outcome measure.
Time Frame: 6-weeks
Population: t-test; missing data for some participants due to attrition or technical difficulties in test administration
Measure: Mean (Standard Deviation); unit: Dollars
Arm/Group | Cognitive Training | Placebo Control
Number analyzed (Participants) | 26 | 28
Dollars | 760.65 (1547.92) | -371.40 (1929.80)

6. Primary Outcome: Trail Making Test (TMT) - Part B
Description: On TMT Part B (Reitan, 1955) participants are asked to connect consecutively numbered and lettered circles, alternating between letters and numbers, as quickly as possible (speeded set-shifting). Test scores were normalized to a t-score with a mean = 50; SD =10; with higher scores indicating better set-shifting abilities.
Time Frame: 6-weeks
Population: T-test; missing data for some participants due to attrition or technical difficulties in test administration
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Training | Placebo Control
Number analyzed (Participants) | 26 | 28
units on a scale | 51.00 (12.71) | 49.93 (11.71)

7. Primary Outcome: The Wisconsin Card Sorting Test - Computer Version 4 Research Edition
Description: The Wisconsin Card Sorting Test - computer version 4 Research Edition (WCST; Heaton et al., 1993) uses stimulus cards to assess set-shifting, an index of cognitive flexibility. Participants must match a stimulus card to the appropriate card deck based on shape designs and rules that shift throughout the task. Scores were normed with t-scores with a mean = 50; SD =10; and higher scores indicating more cognitive flexibility.
Time Frame: 6-weeks
Population: t-test; missing data for some participants due to attrition or technical difficulties in test administration
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Training | Placebo Control
Number analyzed (Participants) | 26 | 28
units on a scale | 48.65 (14.25) | 51.38 (7.28)

8. Primary Outcome: The Tower Test (DKEFS)
Description: The Tower Test is included in the Delis-Kaplan Executive Function System Tests (DKEFS; Delis et al., 2001) and participants are tasked with moving five disks across three pegs to construct a target tower in the fewest number of moves possible. The Tower test will be used to assess planning and procedural problem solving. Scores were normed to a standardized score with a mean = 10; SD =3; with higher scores indicating better problem solving abilities.
Time Frame: 6-weeks
Population: t-test; missing data for some participants due to attrition or technical difficulties in test administration
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Training | Placebo Control
Number analyzed (Participants) | 26 | 28
units on a scale | 11.83 (1.97) | 11.00 (2.00)

9. Secondary Outcome: Functional Status - Inventory of Psychosocial Functioning
Description: The 80-item Inventory of Psychosocial Functioning (IPF; Marx et al., 2009), was developed among Veterans to assess level of functional impairment. The IPF includes 80 self-report and behavioral indices that assess current psychosocial functioning across 7 domains. Domain scores are summed to yield a total score for psychosocial functioning. The IPF yields a grand mean and seven subscale means for functioning in romantic partnerships, family, friendships, parenting, education, work, and self-care activities. Items are rated from 0 (never) to 6 (always). Each subscale is scored by summing scored items, dividing by the maximum possible score, and multiplying by 100, yielding grand and subscales means of 0-100, with higher scores indicating greater impairment. Because participants may skip subscales that do not apply (except for the self-care subscale), the sum of the IPF subscale means is divided by the number of subscales completed.
Time Frame: 6-weeks
Population: t-test; missing data for some participants due to attrition or technical difficulties in test administration
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Control Group: This group will receive 22.5 hours of placebo cognitive training over the course of 6 weeks.
Arm/Group | Cognitive Training | Control Group
Number analyzed (Participants) | 26 | 28
units on a scale | 40.41 (13.53) | 40.94 (11.12)

10. Secondary Outcome: PTSD Symptom Severity
Description: The PTSD Checklist - Military Version (PCL-M; Weathers et al., 2012; National Center for PTSD) is comprised of 20 items that correspond to the 20 DSM-5 (APA, 2013) symptoms of PTSD. The PCL-M provides an index of global PTSD symptom severity and will be administered throughout the study. Scores can range from 0-80 with higher scores indicating higher levels of PTSD symptom severity.
Time Frame: 6-weeks
Population: t-test; missing data for some participants due to attrition or technical difficulties in test administration
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Training | Placebo Control
Number analyzed (Participants) | 26 | 28
units on a scale | 36.04 (16.15) | 40.64 (19.59)

ADVERSE EVENTS:
Time Frame: 5-6 months
Arm/Group | Cognitive Training | Placebo Control
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/38
Other Adverse Events (participants affected / at risk) | 0/52 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan: cover page (2014-06-01): https://cdn.clinicaltrials.gov/large-docs/79/NCT02929979/Prot_SAP_000.pdf